CLINICAL TRIAL: NCT03645109
Title: Effect of Suplementation of 5,000 UI Vitamin D3 on the Glycemic Profile in Patients With Gestational Diabetes Mellitus of the Hospital Civil de Guadalajara Dr. Juan I. Menchaca
Brief Title: Effect of Suplementation of Vitamin D in Gestational Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eva Elizabet Camarena Pulido (Other)
Responsible Party: Sponsor-Investigator, Eva Elizabet Camarena Pulido, Clinical professor, Hospital Civil Juan I. Menchaca
Organization: Hospital Civil Juan I. Menchaca (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0240/18HCJIM/18
Record Dates: First submitted 2018-08-22; First posted 2018-08-24 (Actual); Last update posted 2021-04-02 (Actual); Status verified 2021-03

CONDITIONS: Vitamin D3; Gestational Diabetes Mellitus in Pregnancy
MeSH Terms: interventions — Cholecalciferol

STUDY DESIGN:
Intervention Model Description: Parallel design, two arms
Who Masked: Participant, Care Provider
Masking Description: The capsules with vitamin D or placebo have the same organoleptic characteristics. The jars and envelopes that contain them are identical. The envelopes are identified by a code that only knows who will analyze the data
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin D (Experimental): Will receive capsules with 5,000 IU of vitamin D3, one capsule orally once a day for eight weeks
  Interventions: Dietary Supplement: Vitamin D3
- Placebo (Placebo Comparator): Will receive capsules with placebo (talcum food grade) one capsule orally once a day for eight weeks
  Interventions: Other: Capsules with placebo (talcum food grade)

INTERVENTIONS:
Dietary Supplement: Vitamin D3 — Capsules with 5,000 IU of vitamin D3 once a day (one capsule)
  Arms: Vitamin D
Other: Capsules with placebo (talcum food grade) — Capsules with placebo (talcum food grade)
  Arms: Placebo

SUMMARY:
Randomized double-blind placebo-controlled clinical trial. Consists of the administration of 5,000 IU of vitamin D3 vs Placebo in patients with gestational diabetes mellitus during eight weeks. The objective is to analyze the effects of the intervention on the biochemical parameters that are part of the glycemic profile (insuline, HBA1c, glucose)

DETAILED DESCRIPTION:
Two groups of patients diagnosed with gestational diabetes mellitus. Once the selection criteria are verified, they will be assigned randomly in one of the two arms,one of them will recive 5,000 IU of vitamin D and the other one placebo (talcum food grade). Baseline measurements of vitamin D, glucose,insulin, HBA1c, calcium, phosphorus. At the end of the eight weeks will be determined again the aforementioned biochemical parameters.

ELIGIBILITY:
Inclusion Criteria: Patients with a single pregnancy.

* Patients diagnosed with GDM, which were diagnosed by a glucose tolerance curve 100 grams of glucose, with two altered results from the following: fasting> 95 miligrams / deciliter, 1 hour> 180miligrams / deciliter, 2 hour> 155miligrams / deciliter, 3hous> 140 miligrams / deciliter.
* Gestational age between 24 -30 weeks confirmed with ultrasound of the 1st or 2nd trimester
* Age between 18 and 40 years.

Exclusion Criteria: Patients with pre-existing diabetes mellitus

* Patients with predictive factors for vitamin D hypovitaminosis such as: use of anticonvulsants, renal disease, glomerular filtration rate <60milliliters / minute, thyroid disease or any other pre-existing endocrinological disorders.
* Hypercalciuria> 300 miligrams / day
* Patients taking vitamin D supplementation during the 6 months prior to the study (does not include polyvitamins with lower vitamin D concentrations <500 IU)
* Active and passive smoking patients.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2020-02-28 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-03-10 (Actual)

PRIMARY OUTCOMES:
Changes in the parameters that make up the glycemic profile | Eight weeks
  Glucose, HBA1c, insuline,

SECONDARY OUTCOMES:
Changes in calcium, phosphorus and vitamin D3 | Eight weeks
  Concentrations of calcium and phosphorus in blood and urine and vitamin D in blood

CONTACTS AND LOCATIONS:
Overall Officials: Salvador Mora, Principal Investigator — OPD Hospital Civil de Guadalajara
Locations (1):
- Eva Elizabet Camarena Pulido, Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hollis BW, Johnson D, Hulsey TC, Ebeling M, Wagner CL. Vitamin D supplementation during pregnancy: double-blind, randomized clinical trial of safety and effectiveness. J Bone Miner Res. 2011 Oct;26(10):2341-57. doi: 10.1002/jbmr.463. Erratum In: J Bone Miner Res. 2011 Dec; 26(12):3001. PMID 21706518
- [Result] Yu CK, Sykes L, Sethi M, Teoh TG, Robinson S. Vitamin D deficiency and supplementation during pregnancy. Clin Endocrinol (Oxf). 2009 May;70(5):685-90. doi: 10.1111/j.1365-2265.2008.03403.x. Epub 2008 Sep 2. PMID 18771564
- [Result] Parildar H, Dogruk Unal A, Aksan Desteli G, Cigerli O, Guvener Demirag N. Frequency of Vitamin D deficiency in pregnant diabetics at Baskent University Hospital, Istanbul. Pak J Med Sci. 2013 Jan;29(1):15-20. doi: 10.12669/pjms.291.2896. PMID 24353500
- [Result] Yazdchi R, Gargari BP, Asghari-Jafarabadi M, Sahhaf F. Effects of vitamin D supplementation on metabolic indices and hs-CRP levels in gestational diabetes mellitus patients: a randomized, double-blinded, placebo-controlled clinical trial. Nutr Res Pract. 2016 Jun;10(3):328-35. doi: 10.4162/nrp.2016.10.3.328. Epub 2016 May 16. PMID 27247730